CLINICAL TRIAL: NCT06196151
Title: The Effect of Antenatal Education on Fear of Birth, Physiological Ability to Give Birth and Traumatic Birth Perception: A Randomised Controlled Study
Brief Title: The Effect of Antenatal Education on Fear of Birth, Physiological Ability to Give Birth and Traumatic Birth Perception
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Sinem Göral Türkcü, Assistant Prof., Assistant Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-60116787-020-462207
Record Dates: First submitted 2023-12-18; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Healthy Volunteers; Pregnancy Trimester, Second; Pregnancy Trimester, Third; Nulliparity
Keywords: Antenatal Education; Fear of Birth; Physiological Ability to Give Birth; Traumatic Birth Perception
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Behavioral: Antenatal training
- No intervention (No Intervention)

INTERVENTIONS:
Behavioral: Antenatal training — Training hours: Training will be completed in a total of three weeks and six hours, two hours each week.
  Method: The training will be given online via Zoom application. The training will consist of a total of three weeks and six hours, two hours each week. "Informed Voluntary Consent Form" will be obtained from individuals in both groups. Pregnant women in both the control and intervention groups will be asked to fill out the "Women's Introductory Information Form". The data of the intervention group will be filled out before the first Antenatal education lesson and after all six-hour Antenatal education lessons are completed. The data of the control group will be filled in parallel with the intervention group.
  Group to receive the training: Healthy pregnant women who are at the 20th gestational week at the earliest will be included in the training. Trainings will be carried out in closed groups.
  Arms: Experimental

SUMMARY:
Today, pregnancy and childbirth are important life events that involve many challenges and changes for both men and women. During this process, changes occur in the pregnant woman's body, emotional state and family life. These changes often lead to anxiety about the health of the baby and her own health and to the creation of new stressful situations. During antenatal education, deep relaxation and breathing techniques taught to pregnant women during labour and delivery allow the mother to relax and cope with birth pains more easily and on her own. There are not enough studies in the literature to evaluate the effectiveness of online antenatal classes. In cases where face-to-face antenatal education is not possible during pregnancy, online education is an important option. In the literature, there is no study evaluating how antenatal education affects women's fear of childbirth, physiological ability to give birth and traumatic birth perception together. Therefore, the aim of this study is to examine the effect of antenatal education on fear of childbirth, physiological ability to give birth and perception of traumatic birth. The type of the study is a randomised controlled experimental study with pre-post and control group. The research will be conducted in the form of online training meetings on pregnant women reached through social media. The population of the study will consist of healthy pregnant women who apply to the researchers as a result of the announcements made through social media and who are at the 20th gestational week at the earliest. The sample size was determined by t-test analysis in independent groups in G*power statistical programme, based on two variables, 0.05 significance level, 80% power and medium effect (0.50). Accordingly, a total of 42 pregnant women, 21 pregnant women in each group, are planned to be included in the study. Intention-to-treat analysis will be performed to prevent bias and losses. As an intervention programme, a total of three weeks and six hours of childbirth preparation training will be given, two hours each week. The programme has been prepared by faculty members who have conducted childbirth preparation classes, based on the literature and by making use of childbirth preparation philosophies and methods.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary acceptance to participate in the research
* Being over 18 years of age
* Being at the 20th gestational week at the earliest.
* Not carrying a high risk in pregnancy
* Nulliparity
* Expected to have a normal spontaneous labour

Exclusion Criteria:

* Refusal to participate in the research
* Failure to complete six hours of the childbirth preparation class
* Inability to use the Zoom application
* Psychiatric illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Being over 18 years of age Being at the 20th gestational week at the earliest
Enrollment: 42 (Estimated)
Dates: Start 2024-01-25 (Estimated); Primary Completion 2024-02-08 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | Baseline (It will be applied before starting the intervention)
  This form, which was developed in line with the literature, consists of 9 questions to obtain some socio-demographic characteristics and obstetric information of pregnant women.
Preparation for Labor and Birth (P-LAB) Instrument | Baseline (It will be applied before starting the intervention)
  The Preparation for Labor and Birth (P-LAB) Instrument was developed by Neerland and colleagues (Neerland et al., 2020). It was conducted to determine the confidence of pregnant women in their physiological ability to give birth. The scale is 5-point Likert type and consists of 22 items. The scale consists of four sub-dimensions. The Turkish validity and reliability study of the scale was conducted by Uludağ and Uçtu (2022). Cronbach's alpha value is above 0.70 for all scales and subscales.
Traumatic Birth Perception Scale | Baseline (It will be applied before starting the intervention)
  The scale developed by Yalnız et al. (2016) to measure the perception of traumatic birth in women (18-40 years old) consists of 13 questions and one sub-dimension. The cronbach alpha value of the scale was found to be 0.89. Each question is scored between 0-10 from none to the most severe. As the score obtained from the scale increases, the level of perception of birth as traumatic increases.
Fear of Childbirth Scale for Pregnant Women and Their Partners | Baseline (It will be applied before starting the intervention)
  The Fear of Birth Scale (FOBS) was developed by Haines et al. in 2011 to measure fear of childbirth. Psychometric analyses in Turkish culture were conducted by Serçekuş Ak, Vardar, & Özkan (2018) and it was determined that the scale is a valid and reliable measurement tool that can be used to determine fear of childbirth on pregnant women and their partners in Turkish society. In the Turkish validity and reliability study of the scale, the cronbach alpha internal consistency coefficient was found to be 0.93.

SECONDARY OUTCOMES:
Preparation for Labor and Birth (P-LAB) Instrument | through study completion, an average of one week.
  The Preparation for Labor and Birth (P-LAB) Instrument was developed by Neerland and colleagues (Neerland et al., 2020). It was conducted to determine the confidence of pregnant women in their physiological ability to give birth. The scale is 5-point Likert type and consists of 22 items. The scale consists of four sub-dimensions. The Turkish validity and reliability study of the scale was conducted by Uludağ and Uçtu (2022). Cronbach's alpha value is above 0.70 for all scales and subscales.
Traumatic Birth Perception Scale | through study completion, an average of one week.
  The scale developed by Yalnız et al. (2016) to measure the perception of traumatic birth in women (18-40 years old) consists of 13 questions and one sub-dimension. The cronbach alpha value of the scale was found to be 0.89. Each question is scored between 0-10 from none to the most severe. As the score obtained from the scale increases, the level of perception of birth as traumatic increases.
Fear of Childbirth Scale for Pregnant Women and Their Partners | through study completion, an average of one week.
  The Fear of Birth Scale (FOBS) was developed by Haines et al. in 2011 to measure fear of childbirth. Psychometric analyses in Turkish culture were conducted by Serçekuş Ak, Vardar, & Özkan (2018) and it was determined that the scale is a valid and reliable measurement tool that can be used to determine fear of childbirth on pregnant women and their partners in Turkish society. In the Turkish validity and reliability study of the scale, the cronbach alpha internal consistency coefficient was found to be 0.93.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University Faculty of Health Sciences, Denizli, Kınıklı, Turkey (Türkiye)